CLINICAL TRIAL: NCT06064045
Title: Enhancing Patient Safety and Quality of Care: Study Protocol for a Simulation-based Team Training Intervention Trial
Brief Title: Using Simulation to Support Staff and Improve Quality of Treatment: An Intervention Project Within Pediatrics
Acronym: PAEDSIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Central Denmark Region (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAEDSIM
Record Dates: First submitted 2023-09-21; First posted 2023-10-03 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2023-09

CONDITIONS: Medical Education; Pediatrics; Patient Outcomes
Keywords: Simulation-based team training; Culture; Sickness absence

STUDY DESIGN:
Intervention Model Description: A controlled intervention study comparing two groups each consisting of four pediatric departments.
  Each group consists of approximately 600 participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): The intervention entails boosting the quantity and frequency of simulation-based team training within the intervention group. Additionally, measures to enhance and support simulation will be introduced within the intervention group.
  Interventions: Behavioral: Simulation-based team training intervention
- Control arm (No Intervention): Performing simulation as usual

INTERVENTIONS:
Behavioral: Simulation-based team training intervention — Participants in the intervention group will aim to participate in simulation at a higher quantity and frequency.
  Moreover, the intervention group:
  1. Enrolled 15 healthcare professionals in a 3-day training program to become simulator facilitators, enabling an increase in the utilization of simulation within the group (October 2022).
  2. Organized a 2-day workshop for all pediatric simulation facilitators with the objective of establishing a more robust and standardized foundation for implementing simulation within their respective departments (March 2023).
  3. Procured essential equipment, including mannequins, SimPads, and monitors (before the intervention period).
  4. Provide simulator facilitators with access to an online repository where they can access scenarios for conducting simulations (during the intervention period).
  Arms: Intervention arm

SUMMARY:
Background:

Effective teamwork and quality care are crucial for patient safety overall. Simulation-based team training offers a valuable approach to improving communication, coordination, and decision-making among healthcare professionals, leading to better outcomes and a safer healthcare environment. By evaluating the effectiveness of this training method, the project aims to contribute to the continuous improvement of healthcare delivery.

Hypothesis: Implementation of simulation-based team training in pediatric departments will lead to improved teamwork, communication, and coordination among healthcare professionals, resulting in enhanced patient outcomes and a safer healthcare environment.

Setup: From April 2023 to April 2024 a simulation-based training program will be implemented. The intervention group consists of healthcare professionals working as physicians or nurses in four pediatric departments. The intervention entails increasing the quantity of simulation-based team training within the intervention group. Additionally, measures to enhance and support simulation will be introduced within the intervention group.

Concurrently, another four pediatric departments will serve as a control group, in which no intervention will be implemented.

Both groups consist of approximately 600 healthcare professionals, contributing to a total of 1,200 participants included in this project.

Data collection:

Registration of simulation: The simulation facilitator responsible for each session completes a brief web-based questionnaire made readily accessible from all platforms by QR-code. Data includes Regional ID (unique personal identifier), gender, age, profession, simulation duration, and content, as well as learning goals.

Outcome measures include 1) patient safety culture, 2) rate of sick leave among healthcare professionals, 3) Apgar score, and 4) an intervention cost-benefit analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Employed in one of the eight included pediatric departments during the project period (April 2022 to April 2023)
2. Profession as doctor or nurse

Exclusion Criteria:

1) If participants are employed in both intervention and control group during the project period

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1238 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Sick leave | Up to 30 months
  Change from before intervention to after intervention assessed by administrative human resources database
Patient safety culture | Up to three months
  Change from baseline to after intervention assessed by SAQ-DK Questionnaire
Apgar score | Up to 30 months
  Change from before intervention to after intervention assessed by administrative human resources database
  The Apgar score is based on a score of 1 to 10, determining how well the baby tolerated the birthing process. The higher the Apgar score, the better the baby is doing after birth

CONTACTS AND LOCATIONS:
Overall Officials: Anders Schram, Principal Investigator — Central Denmark Region
Locations (1):
- Corporate HR, MidtSim, Central Denmark Region, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schram AL, Bonne NL, Henriksen TB, Hertel NT, Lindhard MS. Factors associated with participation in simulation-based training. Dan Med J. 2025 Jun 12;72(7):A12240914. doi: 10.61409/A12240914. PMID 40600675
- [Derived] Schram A, Bonne NL, Henriksen TB, Paltved C, Hertel NT, Lindhard MS. Simulation-based team training for healthcare professionals in pediatric departments: study protocol for a nonrandomized controlled trial. BMC Med Educ. 2024 Jun 1;24(1):607. doi: 10.1186/s12909-024-05602-z. PMID 38824537